CLINICAL TRIAL: NCT00162019
Title: Phase 3, Prospective, Multicenter Study to Evaluate the Pharmacokinetics, Immunogenicity, Safety, and Efficacy of IMMUNATE Solvent Detergent (IMMUNATE SD) in Previously Treated Patients With Severe or Moderately Severe Hemophilia A
Brief Title: Pharmacokinetics, Efficacy and Safety Study of IMMUNATE SD (Human Plasma-Derived Coagulation Factor VIII Concentrate) in Hemophilia A Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 040201
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Human Plasma-Derived Coagulation Factor VIII Concentrate (Virus Inactivated by Polysorbate 80 Treatment and Vapor Heat Treatment)

SUMMARY:
The purpose of this study is to evaluate whether IMMUNATE S/D is effective and safe in the treatment of hemophilia A patients. The study consists of 3 parts: Part 1 is a pharmacokinetic comparison of IMMUNATE S/D and its predecessor IMMUNATE. Part 2 is an evaluation of efficacy and safety of IMMUNATE S/D. Part 3 is a pharmacokinetic study of IMMUNATE S/D.

ELIGIBILITY:
Inclusion Criteria:

- Plasma factor VIII level as follows: for Parts 1 & 3: Subjects with severe hemophilia A (plasma baseline factor VIII level <= 1% measured at time of screening) for Part 2: Subjects with severe (plasma baseline factor VIII level <= 1% measured at time of screening) or moderately severe hemophilia A (plasma baseline factor VIII level <= 2% measured at time of screening)

* Males >= 12 but <= 65 years of age
* >= 35 kg body weight
* Previously treated with factor VIII concentrate(s) for a minimum of 150 exposure days (as documented in the subject's medical history)
* Evidence of a protective titer to HAV and HBV at the time of screening
* Immunocompetent as defined by a CD4+ lymphocyte count >400/mm3 and an absolute neutrophil count (ANC) >1500
* Signed informed consent obtained from subject or legally authorized representative

Exclusion Criteria:

* Documented history of inhibitor to factor VIII with a titer >= 0.8 BU
* Current evidence of inhibitor to factor VIII with a titer >= 0.8 BU, measured at the time of screening
* Abnormal renal function (serum creatinine > 1.5 mg/dL)
* HIV-seropositive individuals with any of the following at the time of screening:
* CD4+ lymphocyte count >400/mm3
* AIDS-related complex
* symptomatic AIDS Note: HIV-seropositive subjects with an absolute CD4+ lymphocyte count > 400/mm3 are eligible to participate. HIV-seropositive subjects receiving highly active anti-retroviral therapy (HAART) regimens are eligible for enrollment if they are not excluded by the above criteria
* Active hepatic disease (ALT and AST levels > 5 times the upper limit of normal)
* Clinical or laboratory evidence of hepatic cirrhosis including (but not limited to) a recent and persistent INR (international normalized ratio) > 1.4, the presence of splenomegaly and/or significant spider angiomata on physical exam, and/or a history of esophageal hemorrhage or documented esophageal varices
* Known hypersensitivity to IMMUNATE
* The subject is currently participating in another investigational drug study, or has participated in any clinical study involving an investigational drug within 30 days of study entry
* The subject is currently receiving, or is scheduled to receive during the course of the study, an immunomodulating drug other than anti-retroviral chemotherapy (e.g., a-interferon, steroids at a dose greater than 10 mg/day)
* The subject is identified by the investigator as being unable or unwilling to perform study procedures

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-03-31 (Actual); Primary Completion 2004-08-24 (Actual); Study Completion 2004-08-24 (Actual)

PRIMARY OUTCOMES:
To compare the PK parameters of IMMUNATE S/D and IMMUNATE in subjects with severe hemophilia A (baseline factor VIII <= 1%) | Within 30 minutes pre-infusion; and at 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 9 hours, 24 hours, 28 hours, 32 hours, and 48 hours post-infusion.
to re-evaluate PK parameters for IMMUNATE S/D after a minimum of 14 weeks ± 7 days of treatment with at least 10 exposure days with IMMUNATE S/D | Within 30 minutes pre-infusion; and at 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 9 hours, 24 hours, 28 hours, 32 hours, and 48 hours post-infusion.
to monitor the incidence of factor VIII inhibitor development over a minimum of 27 weeks ± 7 days or at least 50 exposure days, whichever occurs first, in all subjects | Post-Infusion for a minimum of 27 weeks ±7 days or at least 50 treatment EDs, whichever occurs first.
to evaluate the hemostatic efficacy of IMMUNATE S/D in the management of acute bleeding episodes and in the perioperative management of surgical prophylaxis, if required, over the same period of treatment | Post-Infusion for a minimum of 27 weeks ±7 days or at least 50 treatment EDs, whichever occurs first.
to assess the clinical safety of IMMUNATE S/D | Throughout the study period of approximately 18 months.
to retrospectively explore the PK parameters of the VWF moiety of IMMUNATE S/D in subjects with severe hemophilia A (baseline factor VIII <= 1%). | Up to approximately 6.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- National Centre of Hematology and Transfusiology, Sofia, Bulgaria
- University Hospital Motol, Prague, Czechia
- National Medical Center, National Hemophilia Center, Budapest, Hungary
- Poland (2):
  - Klinika Hemetologii I Onkologii Dzieciecej, Warsaw
  - Klinika Hematologii i Onkologii Dzieciecej, Wroclaw